CLINICAL TRIAL: NCT00277420
Title: A Randomized Controlled Trial of a Culturally-Appropriate Weight Loss Intervention for Overweight Latino Children
Brief Title: Trial of a Culturally-Appropriate Weight Loss Intervention for Overweight Latino Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left institution after losing funding for this PI-initiated study
Sponsor: Medical College of Wisconsin (Other)
Collaborators: United Community Center (Other); Milwaukee SCORES (Unknown); Milwaukee Kickers Soccer Club (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #CHW 05/75, HRRC 214-05
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

INTERVENTIONS:
Behavioral: Comprehensive weight management

SUMMARY:
This project aims to conduct a unique, community-based intervention consisting of a randomized trial of a culturally-appropriate weight loss intervention for overweight Latino children in Milwaukee. The intervention promotes lifestyle changes through a low weight loss regimen, one or more physical activities ranging from soccer to hip-hop dance, and dietary counseling including cooking classes for parents. In addition to weight reduction for overweight Latino children, the project has the potential to reduce missed school days and improve self-esteem and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children must be of Latino descent
* At risk for becoming overweight or is overweight
* 6-17 years old.

Exclusion Criteria:

* Age > 17 years old
* Not overweight or at risk for becoming overweight
* Non-Latino ethnicity/race.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
change in body mass index (BMI) z-score

SECONDARY OUTCOMES:
height, weight, and BMI
percent body fat
physical activity
sedentary activity
dietary habits
the child's quality of life
self-esteem
physical fitness
selected health and use of health services measures (missed school days, parental missed work days, and number of healthcare provider visits for illness by child)
the parents' BMI
the child's satisfaction with opportunities to lose weight and increase physical activity in the past year
the parents' satisfaction with opportunities for the child to lose weight and increase physical activity in the past year
costs

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Flores, MD, Study Director — Center for Advancement of Underserved Children (CAUC), Department of Pediatrics, Medical College of Wisconsin; Jane Brotanek, MD, Principal Investigator — Assistant Professor of Pediatrics, Department of Pediatrics, Medical College of Wisconsin; Julio C Maldonado, BA, Principal Investigator — Project Coordinator II, Center for Advancement of Underserved Children (CAUC), Department of Pediatrics, Medical College of Wisconsin
Locations (1):
- Center for Advancement of Underserved Children (CAUC), Department of Pediatrics, Medical College of Wisconsin, Milwaukee, Wisconsin, United States